CLINICAL TRIAL: NCT06976047
Title: Effectiveness of Visual and Sensory Distraction Tools on Anxiety and Behavior Management in Pediatric Dental Patient
Brief Title: Sensory Distraction Tools on Anxiety Management in Pediatric Dental Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UDDS-Pedo-1-2025
Record Dates: First submitted 2025-05-09; First posted 2025-05-16 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Anaesthesia; Anxiety; Children
Keywords: Behavior Management; Distraction techniques; Pain
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Tell-Show-Do Technique (Other): Evaluation of Tell-Show-Do Technique in the management of anxious pediatric patients during inferior alveolar nerve.
  Interventions: Behavioral: Tell-Show-Do
- Visual distraction using magic tricks (Experimental): Evaluation of Visual distraction using magic tricks in the management of anxious pediatric patients during inferior alveolar nerve.
  Interventions: Behavioral: Visual distraction
- Sensory distraction using sensory toys (Experimental): Evaluation of Sensory distraction using sensory toys in the management of anxious pediatric patients during inferior alveolar nerve.
  Interventions: Behavioral: Sensory distraction
- Combining visual distraction using magic tricks with sensory distraction using sensory toys (Experimental): Evaluation of combining visual distraction using magic tricks with sensory distraction using sensory toys in the management of anxious pediatric patients during inferior alveolar nerve.
  Interventions: Behavioral: Visual and sensory distraction

INTERVENTIONS:
Behavioral: Tell-Show-Do — The inferior alveolar nerve block will be administered utilizing a combination of the Tell-Show-Do technique and verbal distraction. Initially, the procedure will be explained to the child in simple, age-appropriate language to reduce fear and foster understanding ("Tell"). This will be followed by a demonstration of the materials and sensations involved, using models or non-threatening demonstrations on the child's hand ("Show"). Once the child appears comfortable, the actual administration of the nerve block ("Do") will proceed exactly as explained, maintaining consistency between the explanation and the action. Throughout the process, verbal distraction will be continuously employed, engaging the child in non-procedural conversation, offering positive reinforcement, and using calming, encouraging language.
  Arms: Tell-Show-Do Technique
Behavioral: Visual distraction — The child's attention will be distracted before anesthesia by asking the child to participate in the activity and attempt to catch the light. The dentist, using a thumb sleeve placed on their finger, will perform various hand movements. The light in the thumb sleeve is controlled by pressing a battery that turns the light on and off. The child is instructed to catch the light, creating the illusion of passing it from one hand to the other and eventually "swallowing" it into the oral cavity. Once the child appears comfortable, the actual administration of the nerve block will proceed.
  Arms: Visual distraction using magic tricks
Behavioral: Sensory distraction — During the application of local anesthesia, the child will be provided with a Pop-it toy as a form of sensory distraction. The child will be briefly instructed on how to use the toy, with a simple explanation of the method of play, encouraging active engagement throughout the anesthetic procedure.
  Arms: Sensory distraction using sensory toys
Behavioral: Visual and sensory distraction — The child's attention will be distracted before anesthesia by asking the child to participate in the activity and attempt to catch the light. The dentist, using a thumb sleeve placed on their finger, will perform various hand movements. The child is instructed to catch the light, creating the illusion of passing it from one hand to the other and eventually "swallowing" it into the oral cavity. During the application of local anesthesia, the child will be provided with a Pop-it toy as a form of sensory distraction. The child will be briefly instructed on how to use the toy, with a simple explanation of the method of play, encouraging active engagement throughout the anesthetic procedure.
  Arms: Combining visual distraction using magic tricks with sensory distraction using sensory toys

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of visual and sensory distraction prior to inferior alveolar nerve block administration in healthy children of both genders, aged 4-6 years.

The main questions it aims to answer are:

* How effective are different visual and sensory distraction techniques in reducing pain and anxiety during inferior alveolar nerve block procedures in young children?
* Which type of distraction technique (visual or sensory) is the most effective? This study will compare children receiving visual and sensory distraction with those receiving no distraction to assess differences in pain perception and anxiety levels during the procedure.

Participants will:

* Undergo a standardized inferior alveolar nerve block procedure.
* Be randomly assigned to one of the following groups: visual distraction, sensory distraction, or control (no distraction).
* Complete simple self-reported pain and anxiety assessments appropriate for their age (such as the Wong-Baker FACES Pain Rating Scale).
* Be evaluated using additional objective measures, including the FLACC scale and heart rate monitoring.

DETAILED DESCRIPTION:
Dental anxiety is considered one of the most common challenges in pediatric dentistry, as it directly affects - and may limit - a child's cooperation during treatment.

Distraction techniques work by diverting the child's attention away from painful or difficult therapeutic procedures and are considered highly important in managing children's behavior within the dental clinic.

Various visual and/or auditory distraction methods can be employed by the dental team when working with pediatric patients. Distraction techniques may be either active (such as allowing the child to play electronic games) or passive (such as listening to music or watching animated movies).

These techniques are considered a valuable alternative to pharmacological preparation for completing dental treatments in children, and many pediatric dentists have adopted them as an effective strategy for managing dental anxiety in young patients.

Despite the availability of numerous behavioral management techniques for addressing dental anxiety, the effectiveness of different distraction methods - whether visual, sensory, or a combination of both - still requires further investigation.

ELIGIBILITY:
Inclusion Criteria:

1. no previous dental experience.
2. definitely positive or positive ratings of Frank scale.
3. Need of IAN block for any dental treatment.

Exclusion Criteria:

1. previous dental experience
2. systematic or mental disorders.
3. definitely negative or negative ratings of Frankel scale
4. Any contraindication for regional anesthesia

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-07-22 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Pain levels | 5 minutes following the inferior alveolar nerve block injection.
  Pain levels will be measured by using a self-reported simplified Wong-Baker faces pain scale: 0 no Hurt - 1 Hurts little Bit - 2 Hurts little More - 3 Hurts Even More - 4 Hurts Whole Lot - 5 Hurts Worst
Anxiety levels | 1 minute during inferior alveolar nerve block administration
  This will be evaluated using the Face-Legs-Activity-Cry-Consolability (FLACC) scale (0 low anxiety and pain level - 10 high anxiety and pain level).

SECONDARY OUTCOMES:
Pulse rate | (1) five minutes after the patient is seated comfortably on the dental chair, (2) five minutes following the injection of the anesthetic drug
  Pulse rate (the number of times your heart beats each minute bpm will be evaluated using Finger Pulse Oximeter.

CONTACTS AND LOCATIONS:
Overall Officials: Alaa M Snobar, DDS, Principal Investigator — Damascus University; Chaza N Kouchaji, PhD, Study Chair — Damascus University
Locations (1):
- School of Dental Medicine, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Su HC, Hsieh CW, Lai NM, Chou PY, Lin PH, Chen KH. Using Vibrating and Cold Device for Pain Relieves in Children: A Systematic Review and Meta-analysis of Randomized Controlled Trials. J Pediatr Nurs. 2021 Nov-Dec;61:23-33. doi: 10.1016/j.pedn.2021.02.027. Epub 2021 Mar 16. PMID 33735633
- [Background] Alsibai E, Bshara N, Alzoubi H, Alsabek L. Assessing an active distracting technique during primary mandibular molar pulpotomy (randomized controlled trial). Clin Exp Dent Res. 2023 Apr;9(2):283-289. doi: 10.1002/cre2.702. Epub 2022 Dec 8. PMID 36478192
- [Background] Kothari P, Mathur A, Chauhan RS, Nankar M, Tirupathi S, Suvarna A. Effectiveness of thaumaturgic distraction in alleviation of anxiety in 4-6-year-old children during inferior alveolar nerve block administration: a randomized controlled trial. J Dent Anesth Pain Med. 2023 Jun;23(3):143-151. doi: 10.17245/jdapm.2023.23.3.143. Epub 2023 May 26. PMID 37313267
- [Background] Hart R, Walton M. Magic as a therapeutic intervention to promote coping in hospitalized pediatric patients. Pediatr Nurs. 2010 Jan-Feb;36(1):11-6; quiz 17. PMID 20361440
- [Background] Bawaeda O, Wanda D, Aprillia Z. Effectiveness of pop-it therapeutic play on children's anxiety during inhalation therapy in children's wards. Pediatr Med Chir. 2023 Mar 28;45(s1). doi: 10.4081/pmc.2023.315. PMID 36974915